CLINICAL TRIAL: NCT05811845
Title: Optimizing the Maintenance Phase of Childhood Acute Lymphoblastic Leukemia AIEOP Protocol Through Mercaptopurine Therapeutic Drug Monitoring and Proactive Strategies for Adherence
Brief Title: Mercaptopurine Therapeutic Drug Monitoring to Optimize the Maintenance Phase of Childhood ALL
Status: Recruiting | Type: Observational
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Sponsor
Other Study IDs: 57/22
Record Dates: First submitted 2023-03-31; First posted 2023-04-13 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Acute lymphoblastic leukemia; Compliance; Mercaptopurine
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Patient Compliance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute lymphoblastic leukemia (ALL) is the most common hematological malignancy in children (<18 years). The success of pediatric ALL therapy is remarkable but important challenges still need to be faced, including cure rates in specific patients' subsets (e.g.: adolescents and relapsed patients), and short- and long-term chemotherapy-related toxicities. The therapeutic scheme of the Associazione Italiana Emato-oncologia pediatrica (AIEOP) ALL protocols consists in a more intensive and toxic earlier phase (to induce and consolidate remission, about 6 months), followed by a prolonged period of immunosuppression (achieved by self- or parent-administered daily mercaptopurine (MP) and weekly methotrexate (MTX) per os). It is now well established that the length of the maintenance phase (up to 24 months after diagnosis) is as necessary as the early remission induction for sustained event-free survival (EFS). Both MP and MTX can lead to potentially serious complications, including potentially life-threatening myelosuppression and infections. To exert its therapeutic effect, MP requires an intracellular enzymatic conversion into active thionucleotides (TGN) and is thus susceptible to intra- and inter-individual variations in efficacy and toxicity. Patients carrying variants in TPMT and NUTD15 genes are at risk of adverse effects when treated with standard MP doses: these patients are identifiable by pre-emptive genotyping. Recent studies demonstrated that an adequate and constant MP exposure during maintenance is associated with higher therapeutic success. Prescribed MP doses are often changed by physicians to target a white blood cell count (WBC) range of 2.0-3.0 × 109/L during maintenance. In the AIEOP ALL 2009 protocol, patients with lower mean TGN exposure during maintenance showed a trend towards a higher risk of relapse compared to others. Similarly, patients with higher intra-individual variability in TGN over time showed a trend towards a worse outcome. Daily compliance to prescribed MP over time is a challenging issue for patients and may result in less effective therapy. The high intra-individual variability in exposure due to the frequent dose adjustments and the potential lack of patients' adherence to oral MP therapy over time might contribute to the risk of relapse. The aim of this study is to assess through therapeutic drug monitoring of MP if patients' exposure during maintenance is adequate and constant.

DETAILED DESCRIPTION:
Acute lymphoblastic leukemia (ALL) is the most common hematological malignancy in children (<18 years). The success of pediatric ALL therapy is remarkable (5 years survival ~90%). However, important challenges still need to be faced, including cure rates in specific patients' subsets (e.g.: adolescents and relapsed patients, 5 years survival ~60-70% and ~40-50%, respectively), and short- and long-term chemotherapy-related toxicities. The therapeutic scheme of the Associazione Italiana Emato-oncologia pediatrica (AIEOP) ALL protocols consists in a more intensive and toxic earlier phase (to induce and consolidate remission, ~ 6 months), followed by a prolonged period of immunosuppression (achieved by self- or parent-administered daily mercaptopurine (MP) and weekly methotrexate (MTX) per os). It is now well established that the length of the maintenance phase (up to 24 months after diagnosis) is as necessary as the early remission induction for sustained event-free survival (EFS). Ideally, the combination of antimetabolites MP and MTX is safe enough to provide the required antileukemic effects with minimal adverse events. However, both drugs can lead to potentially serious complications, including potentially life-threatening myelosuppression and infections. To exert its therapeutic effect, MP requires an intracellular enzymatic conversion into active thionucleotides (TGN) and is thus susceptible to intra- and inter-individual variations in efficacy and toxicity. In particular, patients carrying variants in TPMT and NUTD15 genes are at risk of adverse effects when treated with standard MP doses: these patients are identifiable by pre-emptive genotyping, and pharmacogenetic-based dose adjustment guidelines are already available. Recent studies of the Children's Oncology Group (COG) and of the Nordic Society of Pediatric Hematology and Oncology (NOPHO) demonstrated that an adequate and constant MP exposure during maintenance is associated with higher therapeutic success. Prescribed MP doses are often changed by physicians to target a white blood cell count (WBC) range of 2.0-3.0 × 109/L during maintenance. In the AIEOP ALL 2009 protocol, patients with lower mean TGN exposure during maintenance (below median cut-off of 272.44 pmol/10x108 RBC) showed a trend towards a higher risk of relapse compared to others (11.5% vs 5.5%, respectively). Similarly, patients with higher intra-individual variability in TGN over time (above the 75th percentile of the coefficient of variation (CV)) showed a trend towards a worse outcome (10.3% vs 4.8%). These preliminary data were obtained in 265 ALL patients (age: median (interquartile range): 4.82 (3.03-8.53) years; 58.5% male; follow up from maintenance beginning: 1338 (1377-4162) days; 27 relapsed, TGN measured in 391 blood samples of 209 patients). Daily compliance to prescribed MP over time is a challenging issue for patients and may result in less effective therapy: indeed, the recent use of an electronic device - the medication bottle cap opening (MEMS)- revealed that patients' self-reported MP intake overestimates true intake, in particular in some sociodemographic groups. Adherence is generally poorer in adolescents compared to younger children, likely because drug administration may no more be under strict parents' supervision: this lower compliance can in part contribute to the survival disparity observed between the two age groups. Thus, the high intra-individual variability in exposure due to the frequent dose adjustments and the potential lack of patients' adherence to oral MP therapy over time might contribute to the risk of relapse.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed ALL
* Age <18 years at diagnosis
* Written informed consent given

Exclusion Criteria:

-

Max Age: 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children with new diagnosis of ALL
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-07-30 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To establish the variability of MP systemic exposure (TGN) over time | After 18 months from the start of treatment
  MP metabolites will be evaluated in erythrocytes of peripheral blood according to standardized methods
To establish the correlation between MP systemic exposure (TGN) and absolute neutrophil count to identify the ideal TGN therapeutic range | After 18 months from the start of treatment
  MP metabolites will be evaluated in erythrocytes of peripheral blood according to standardized methods
To establish if TGN levels and intra-individual variability (TGN-CV) could monitor patients' adherence during the long-term maintenance phase | After 18 months from the start of treatment
  MP metabolites will be evaluated in erythrocytes of peripheral blood according to standardized methods
To determine the impact of TGN on EFS | After 18 months from the start of treatment
  MP metabolites will be evaluated in erythrocytes of peripheral blood according to standardized methods

CONTACTS AND LOCATIONS:
Overall Officials: Marco Rabusin, MD, Study Director — IRCCS materno infantile Burlo Garofolo
Locations (4):
- Italy (4):
  - Fondazione MBBM / A.O. San Gerardo, Monza, Monza Brianza
  - IRCCS Ospedale Pediatrico "Bambino Gesù", Roma
  - Presidio Infantile Regina Margherita, Torino
  - IRCCS materno infantile Burlo Garofolo, Trieste

IPD SHARING:
Plan to Share IPD: No